CLINICAL TRIAL: NCT00104988
Title: A Phase II Trial of Combination Thalidomide Plus Temozolomide in Patients With Metastatic Malignant Melanoma
Brief Title: S0508: Thalidomide and Temozolomide in Treating Patients With Stage IV Melanoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000412048; S0508 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Temozolomide; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thalidomide and Temozolomide (Experimental): Patients receive oral thalidomide once daily on days 1-56 and temozolomide once daily on days 1-42. Courses repeat every 56 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temozolomide; Drug: thalidomide

INTERVENTIONS:
Drug: temozolomide — 75 mg/m^2/day PO daily for 6 weeks followed by a 2-week break
Drug: thalidomide — 200 mg/day PO daily

SUMMARY:
RATIONALE: Thalidomide may stop the growth of melanoma by blocking blood flow to the tumor. It may also stimulate the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving thalidomide together with temozolomide may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving thalidomide together with temozolomide works in treating patients with stage IV melanoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 6-month progression-free survival of patients with unresectable stage IV malignant cutaneous melanoma treated with thalidomide and temozolomide.
* Determine the objective response (confirmed and unconfirmed complete response and partial response) in patients with measurable disease treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral thalidomide once daily on days 1-56 and temozolomide once daily on days 1-42. Courses repeat every 56 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at week 9, every 2 months until disease progression, and then every 6 months until 3 years from study entry.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study within 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant cutaneous melanoma

  * Unresectable, stage IV disease
  * Unknown primary allowed
* Measurable or non-measurable disease

  * If all known sites of disease are within a previously irradiated port, disease progression must be clearly demonstrated
* No brain metastases by CT scan or MRI within the past 42 days

  * Prior brain metastasis allowed provided both of the following criteria are met:

    * Completely resected and free of disease
    * Treated with whole brain radiotherapy and completed treatment at least 28 days ago

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (transfusions allowed)

Hepatic

* Bilirubin ≤ 3 times upper limit of normal (ULN)
* SGOT or SGPT ≤ 2.5 times ULN (5 times ULN if liver metastases are present)

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception for 4 weeks before, during, and for 4 weeks after study participation
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission
* No history of allergic reaction to dacarbazine

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior thalidomide for stage IV disease
* At least 28 days since prior biological therapy
* At least 28 days since prior immunotherapy
* At least 28 days since prior adjuvant interferon alfa

Chemotherapy

* No prior temozolomide or dacarbazine for stage IV disease
* At least 28 days since prior chemotherapy

Endocrine therapy

* At least 28 days since prior hormonal therapy

Radiotherapy

* See Disease Characteristics
* At least 28 days since prior radiotherapy

Surgery

* See Disease Characteristics
* At least 28 days since prior surgery for primary and stage IV disease

Other

* No more than 1 prior systemic therapy regimen for stage IV disease
* At least 28 days since other prior systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-06; Primary Completion 2007-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 6 months | 6 months after registration
Objective response (confirmed and unconfirmed complete and partial responses) | Week 9, every 8 weeks thereafter until progression
6-month overall survival | six months after registration

CONTACTS AND LOCATIONS:
Overall Officials: Joseph I. Clark, MD, Study Chair — Loyola University; Laura F. Hutchins, MD, Principal Investigator — University of Arkansas
Locations (132):
- United States (132):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Eden Medical Center, Castro Valley, California
  - North Bay Cancer Center, Fairfield, California
  - Saint Rose Hospital, Hayward, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Highland General Hospital at St. George's University School of Medicine, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Christus Schumpert Cancer Treatment Center, Shreveport, Louisiana
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Ted B. Wahby Cancer Center at Mount Clemens General Hospital, Mount Clemens, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Highland Hospital of Rochester, Rochester, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - U.T. Cancer Institute at University of Tennessee Medical Center, Knoxville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Clark JI, Moon J, Hutchins LF, Sosman JA, Kast WM, Da Silva DM, Liu PY, Thompson JA, Flaherty LE, Sondak VK. Phase 2 trial of combination thalidomide plus temozolomide in patients with metastatic malignant melanoma: Southwest Oncology Group S0508. Cancer. 2010 Jan 15;116(2):424-31. doi: 10.1002/cncr.24739. PMID 19918923